CLINICAL TRIAL: NCT05221359
Title: An Open Label, Monocentric, Pilot Study Evaluating Safety of ExOlin® in Patients With Poorly Controlled Type 1 Diabetes With High Glucose Fluctuations, Prone to Severe Hypoglycemia
Brief Title: Pilot Study Evaluating Safety of ExOlin® in Patients With Poorly Controlled Type 1 Diabetes
Acronym: Pilot'Ex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defymed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEXN-T1D-2017-01; 2020-A01763-36 (Registry Identifier: ID-RCB France); 2020-003020-17 (EudraCT Number)
Record Dates: First submitted 2021-12-03; First posted 2022-02-03 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes; Type 1 Diabetes Mellitus With Hypoglycemia
Keywords: Safety; Pilot; Type 1 Diabetes; High glucose fluctuations; Severe Hypoglycemia; Hypoglycemia unawareness; Extraperitoneal; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: All patients enrolled will undergo period with subcutaneous delivery of insulin, as a baseline data collection. Then, patients will receive the ExOlin device, undergo post-implantation FU, and then get insulin therapy via ExOlin. Explantation of the device, when required, will be accompanied by a safety FU.
  During all study phases, NovoRapid insulin will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test arm (Experimental): All patients will be enrolled in same arm which contains the two interventions (device + drug) and follow mandatory phases of trial: screening, implantation, treatment with ExOlin, explantation.
  Interventions: Device: ExOlin®; Drug: Insulin aspart

INTERVENTIONS:
Device: ExOlin® — Implantation of ExOlin® device, safety follow-up followed by a treatment period in which device is used to administer insulin.
  Device explanted with a safety follow-up.
Drug: Insulin aspart — Use of NovoRapid insulin during all periods of the clinical investigations

SUMMARY:
First in Human, pilot investigation An Open Label, Monocentric, Pilot Study Evaluating Safety of ExOlin® in Patients with Poorly Controlled Type 1 Diabetes with High Glucose Fluctuations, Prone to Severe Hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women (age ≥ 18 years);
2. Diagnosis of Type 1 Diabetes (T1D) for more than 2 years at the start of screening;
3. Body mass index (BMI) > 16 kg/m2 and < 35 kg/m2;
4. Well managed intensive SubCutaneous (SC) insulin therapy, i.e. patient using for at least 3 months:

   * CSII, whatever the insulin pump used, and
   * Continuous Glucose Monitoring (CGM), by using Dexcom G6;
5. 7.0% < Serum HbA1c < 12.0%;
6. Patient characterized by one of the following conditions:

   * Unstable diabetes/poor glycemic control, meaning patient presenting:

     * at least one episode of severe hypoglycemia during the 12 months prior to study screening. Severe hypoglycemia is defined by American Diabetes Association (ADA) standards as "severe cognitive impairment requiring assistance from another person for recovery" (as per ADA's definition in "standards of care in diabetes");
     * or glycemic excursions (post-prandial hyperglycemic or nocturnal hypoglycemic episodes) considered as too frequent and of high amplitude by the investigator, during the previous month;
   * Presence of adverse side effects of SC insulin-therapy:

     * SC insulin resistance;
     * or severe acquired lipodystrophy resistant to pump treatment;
     * or genetic skin atrophy or lipodystrophy.

Exclusion Criteria:

1. Renal glomerular filtration rate <30 mL/min/1.73m2 as per Chronic Kidney Disease - Epidemiology Collaboration (CDK-EPI) calculation;
2. Immunocompromised patient;
3. Local or systemic acute or chronic inflammation (rheumatoid arthritis, sclerodermia);
4. Active infection or inflammation;
5. Known history of skin affliction that could impact ExOlin® tolerance;
6. Ongoing active anticoagulant therapy;
7. Severe wound healing issues;
8. Parietal reinforcement prostheses;
9. Known allergy to one of the devices' components, including known allergy to fixation systems (e.g. patch, plaster) for SC administration devices such as external pumps and CGM, or chronic allergy related to prolonged wearing of such systems;
10. Known allergy to insulin NovoRapid®;
11. Known allergy to anesthetics, or products containing iodine and its derivates, or antibiotics used during surgery (cefazolin, and combination of clindamycin and gentamycin);
12. Activity contraindicated as per external pump and CGM use recommendations;
13. Patient willing to practice activities with risks of trauma or major change in the environment pressure such as combat sport or scuba diving;
14. Cardiac condition incompatible with surgery requirements as per anesthesiologist's opinion;
15. Unstable diabetic retinopathy (as per ophthalmologist's review within 6 months before screening);
16. Current or history of unresolved malignancy within 5 years before screening (with exceptions for squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or breast carcinoma without lymph node metastases, well-differentiated thyroid carcinoma or other non-invasive lesion that, in the opinion of the investigator, is considered as cured with minimal risk of recurrence within 5 years);
17. Other surgical or medical condition that, in the judgment of the investigator, might warrant exclusion or be contraindicated, like for instance visual or hand-use symptoms;
18. Mental handicap or psychiatric condition incompatible with appropriate handling of devices or compliance to treatment or investigation-related tasks;
19. Known active alcohol or drug abuse;
20. Having received corticoid treatment within 4 weeks prior to enrollment;
21. Having received an investigational product within 12 weeks prior to enrollment, or currently participating in another clinical trial, with the exception of observational / non-interventional; registries, for which written prior approval of Defymed is needed;
22. Women planning for pregnancy, being pregnant or breastfeeding or unwilling to use adequate contraceptive methods for the duration of the study (oral hormonal contraceptives, implants, injectables, hormonal or copper intrauterine device, or vasectomized partner);
23. Person under guardianship, trusteeship or deprived of liberty;
24. Person not affiliated to one of the French social security systems;
25. Unwilling to give written informed consent to participation in the study, or unable to do so for psychiatric, cognitive or linguistic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety: Percentage of patients who will experience at least one relevant adverse event (AE) judged by the investigator as probably or highly probably related to ExOlin® for the duration of mandatory phases of the study | From implantation of the device (4 weeks after screening visit) till end of post-explantation safety follow-up (week 36), meaning a duration of 32 weeks.
  Percentage of patients who will experience at least one relevant adverse event (AE) judged by the investigator as probably or highly probably related to ExOlin® for the duration of the study :
  * Linked to implantation (any unexpected or severe signs of cutaneous or extraperitoneal intolerance s.a. redness, edema or delayed healing, as per clinical exam of the skin and palpation in regard of the scar and SC port, associated to systemic signs s.a. fever, chills, abnormal biologic values [including: complete blood count, C-reactive protein]);
  * linked to therapeutic use of ExOlin (i.e. to administrate insulin: ExOlin® device failure or local infection);
  * other unexpected related AEs.
  The primary endpoint will be achieved when the device has been retrieved from all enrolled patients and post-explantation observation time (3 months post explantation) has been completed.
Safety: Percentage of patients who will experience at least one relevant adverse event (AE) judged by the investigator as probably or highly probably related to ExOlin® for the whole duration of the study (extension phase included) | From implantation of the device (4 weeks after screening visit) till end of post-explantation safety follow-up, meaning a duration up to of 168 weeks maximum for patients completing extension phase.
  Percentage of patients who will experience at least one relevant adverse event (AE) judged by the investigator as probably or highly probably related to ExOlin® for the duration of the study :
  * Linked to implantation (any unexpected or severe signs of cutaneous or extraperitoneal intolerance s.a. redness, edema or delayed healing, as per clinical exam of the skin and palpation in regard of the scar and SC port, associated to systemic signs s.a. fever, chills, abnormal biologic values [including: complete blood count, C-reactive protein]);
  * linked to therapeutic use of ExOlin (i.e. to administrate insulin: ExOlin® device failure or local infection);
  * other unexpected related AEs.
  The primary endpoint will be achieved when the device has been retrieved from all enrolled patients and post-explantation observation time (3 months post explantation) has been completed.

SECONDARY OUTCOMES:
Safety : Percentage of patients who will experience at least one AE, according to its severity, seriousness, relation with the device or the surgery or the treatment, outcome, by system-organ-class and preferred term. | From implantation of the device through study completion, meaning from 1 month after screening, duration of 8 months for mandatory phases and up to 3 years and 3 months for patients reaching end of extension phase
  Percentage of patients who will experience at least one AE, according to its severity, seriousness, relation with the device or the surgery or the treatment, outcome, by system-organ-class and preferred term.
Safety: Percentage of participants with abnormal vital signs or physical findings. | From implantation of the device through study completion, meaning from 1 month after screening, duration of 8 months for mandatory phases and up to 3 years and 3 months for patients reaching end of extension phase
  Percentage of participants with abnormal vital signs (blood pressures, heart rate, body temperature) or physical findings (i.e. significant abnormal lab results s.a. WBC or observation of abnormal scar)
Early Performance: Glycemic control | 2nd month of treatment (meaning week 20) vs end of screening (week 4)
  Glycemic control as measured by use of a Continuous Glucose Monitor (Dexcom G6): comparison of data collected when ExOlin® is used versus data collected during Continuous Subcutaneous Insulin Infusion (CSII)
Early Performance: Glycemic control | 3rd month of treatment (meaning week 24) vs end of screening (week 4)
  Glycemic control as measured by use of a Continuous Glucose Monitor (Dexcom G6): comparison of data collected when ExOlin® is used versus data collected during Continuous Subcutaneous Insulin Infusion (CSII)
Early Performance: Glycemic control | Every 4 weeks starting from 2nd month of treatment (meaning week 20) and till end of use of ExOlin (up to week 160) vs end of screening (week 4)
  Glycemic control during the global Follow-Up (FU) of the patient across all study (monthly values, by use of Continuous Glucose Monitor Dexcom G6) by comparison of data collected when ExOlin® is used versus data collected during CSII
Early Performance | Baseline, then every 12 weeks up to end of use of ExOlin (up to week 160)
  Glycemic control as per HbA1c
Quality of Life: Overall score and subscores of the Diabetes Quality of Life (DQOL) questionnaire | at the end of the Treatment phase (3rd month of treatment) versus data at the end of the Screening phase (1 month duration)
  Overall score and subscores of the Diabetes Quality of Life (DQOL) questionnaire: scale from 0 to 100. The higher patient rates, the better the outcome is.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France